CLINICAL TRIAL: NCT03193268
Title: Effects of Intensity-matched Agility and Cycling Exercise Training on PD Patients' Clinical Symptoms, Posture, and Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Principal Investoigator, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB0014/2015
Record Dates: First submitted 2017-06-01; First posted 2017-06-20 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2017-07

CONDITIONS: Parkinson Disease; Balance; Rehabilitation; Motor Function
Keywords: sensorimotor training; quality of life; posture
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity agility group (Experimental): Exercise therapy
  Interventions: Other: Single-blind RTC of PD patients
- Non-agility cycling group (Experimental): Parkinson's Bicycle Group, which takes 1 hour of exercise every day for 5 weeks
  Interventions: Other: cycling
- No-exercise control group (No Intervention): Control Parkinson's disease control group thad will not receive exercise treatment

INTERVENTIONS:
Other: Single-blind RTC of PD patients — The groups participate in observation for 5 weeks. Two groups take part in a motion therapy over the 5-week period.
  Arms: High intensity agility group
Other: cycling — Patients must undergo a daily exercise cycle of 1 hour during the intervention
  Arms: Non-agility cycling group

SUMMARY:
Determine the short-term and lasting effects of intensity-matched exercise programs on level 2-3 PD patients' clinical symptoms, postural control, and mobility.

Hypothesis

1. The inclusion of a Borg-scale/heart-rate matched active control group will allow us to test the idea that, in addition to a fitness element, the reflexive movements that chellenge PD patients' sensorimotor system will improve patients' clinical symptoms, posture, and mobility more than fitness training and that such lasting effects will be superior in the agility compared with the fitness-control group. This hypothesis emered from the idea that the favorable results in the currently under review paper may be in part due to a simple conditioning effect instead of a specific motor learning effect caused by the xbox training.
2. If feasible, i.e., if there is a lerge enough pool of patients to randomize, a balance training group will be also added to test the idea that the reflexive actions evoked by the agility program by xbox exergaming still produce superior adaptations vs. the balance group because xbox forces patients to rapidly and reflexively execute movements (respond to cues, prompts), while balance training allows patients to stop, go, stop, and go and disrupt the continous execution of linked movements. The disruptions of movement chains could arise from small losses of balance on the unstabel surfaces, need for patients to re-initiate every movement element of a sequence, planning each movement element. It is not clear yet how it woul be possible to match all three intervention groups on Borg/heart rate intensity.

DETAILED DESCRIPTION:
Agility: Xbox based high intensity program, as detailed in the submitted manuscript. Borg scale after after each exercise block is recorded. Heart rate continuosly measured. These data are used to set intensity in the fitness group.

Fitness: A stationary bicycle ergometer program that includes visual stimulation in the form of watching nature programs and movies to account for visual stimulus in Agility group. Mean heart rate and Borg scale readings from Agility group will form the target intensity.

Control: No-exercise, measurment-only control group.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease,
* Hoenh Yahr scale of 2-3,
* instability problem,

Exclusion Criteria:

• Severe heart problems, severe demeanor, alcoholism, drug problems,

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
EQ5D-5L | 0-5 scale (5 weeks-long, the higher score is better)
  Questionnaire
Borg test | 0-40 point (5 week-long, higher score is better)
  Fatigue questionnaire
PDQ-39 | 0-39 scale (5week-long, higher score is better)
  special Parkinson's Disease test - motor and no-motor function
SPPB test (gait, balance, leg stregth) | 0-12 scale (5 week-long, higher score is better)
  Walking and balance testing

CONTACTS AND LOCATIONS:
Locations (1):
- Somogy Megyei Kaposi Mór Teaching Hospital, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- See also: Description Related Info — https://www.ncbi.nlm.nih.gov/pubmed/